CLINICAL TRIAL: NCT01824095
Title: Chiropractic Care and a Specific Regimen of Nutritional Supplementation for Patients With Acute Ankle Sprain: a Multisite Randomized Controlled Trial
Brief Title: Chiropractic Care and a Specific Regimen of Nutritional Supplementation for Patients With Acute Ankle Sprain
Acronym: ASP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to recruit enough subjects to attain the minimum sample size.
Sponsor: Logan University, Inc. (Other)
Collaborators: Sport and Spine Rehab Clinical Research Foundation (Other); Parker University (Other); Brentwood Spine Clinic, Brentwood, MO, USA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Standard Process - 2013
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Ankle Sprains
MeSH Terms: conditions — Ankle Injuries | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Acute phase (1st treatment through Week 4): Placebo. 2 capsules 3 x day. Chronic phase (Weeks 5-16): Placebo. 1 capsule 3 x day.
  Interventions: Dietary Supplement: Dietary supplement
- dietary supplement (Experimental): Acute phase (1st treatment through Week 4): Ligaplex 1. Ligaplex 1 supplies nutrients to support connective tissue and reduce inflammation. The protocol is commonly used in chiropractic practice and suggested by Standard Process: 2 capsules 3 x day.
  Chronic phase (Weeks 5-16): Glucosamine Synergy. This supplement maintains connective tissue and joint health. The protocol is commonly used in chiropractic practice and suggested by Standard Process: 1 capsule 3 x day.
  Interventions: Dietary Supplement: Dietary supplement

INTERVENTIONS:
Dietary Supplement: Dietary supplement

SUMMARY:
The purpose of this multisite randomized controlled trial (RCT) is to compare the short-term (6 week) and long-term (6 month) effect of chiropractic care combined with a specific nutritional supplement regimen to chiropractic care with a placebo supplement for patients with ankle sprains, in terms of improvement in physical function and pain.

DETAILED DESCRIPTION:
Specific Aim 1: to compare the short-term (6 week) effect of chiropractic care combined with a specific nutritional supplement regimen to chiropractic care with a placebo nutritional supplement for patients with ankle sprains, in terms of speed and amount of improvement in physical function and pain. Our hypothesis is that chiropractic care plus nutritional supplements designed to supply necessary nutrients for ligament healing will have improved outcomes in pain and disability, compared to chiropractic care plus placebo. We will use the Foot and Ankle Ability Measure Activities of Daily Living Subscale (FAAM ADLS) to measure outcomes.

Specific aim 2: to compare the long-term (6 month) effect of chiropractic care combined with a specific nutritional supplement regimen to chiropractic care with a placebo nutritional supplement for patients with ankle sprains, in terms of speed and amount of improvement in physical function and pain. Our hypothesis is that chiropractic care plus nutritional supplements designed to supply necessary nutrients for ligament healing will have improved outcomes as measured by the FAAM ADLS, compared to chiropractic care plus placebo.

Specific aim 3: to explore any changes in the attitude, knowledge and behavior of chiropractic interns and practitioners of the role of nutrition in treating musculoskeletal injuries, pre- and post-intervention. We will also compare their responses to those of a population of students and practitioners who did not participate in the project, as a comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Acute ankle sprain, defined as ankle sprain within the past 7 days, by patient report. Treating clinician will verify diagnosis via clinical examination.
* Ages 18-50; ankle sprains are more common in this age group.

Exclusion Criteria:

* Diagnosis of grade III ankle sprain, fracture or dislocation; fracture will be diagnosed using the Ottawa ankle rules11,12
* Contraindications to chiropractic care, such as fracture or other abnormalities found by history, examination, or x-rays, as determined by the treating or supervising clinician.
* Pregnancy: although it is unlikely that the nutritional supplements would have adverse effects on the fetus, we are excluding pregnant women as a safeguard.
* Unwilling or unable to regularly take the supplements (e.g., vegetarians; known sensitivity by self-report; patients will be shown the ingredient list prior to signing the informed consent).
* Litigation for a health-related claim (in process or pending).
* History of ankle surgery or presence of ankle hardware (pins, screws, etc.), by patient report.
* History of diabetic or other peripheral neuropathy, by patient report.
* Current use of prescription or nonprescription medications that may interact with experimental or placebo supplements, by patient report.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) Activities of Daily Living Subscale (ADLS) | baseline to 6 weeks

SECONDARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) Activities of Daily Living Subscale (ADLS) | baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl K Hawk, DC, PhD, Principal Investigator — Logan University
Locations (9):
- United States (9):
  - Sport and Spine Rehab, Columbia, Maryland
  - Sport and Spine Rehab, Ft. Washington, Maryland
  - Sport and Spine Rehab, Landover, Maryland
  - Sport and Spine Rehab, Rockville, Maryland
  - Brentwood Spine Clinic, Brentwood, Missouri
  - Logan University, Chesterfield, Missouri
  - Sport and Spine Rehab, Fairfax, Virginia
  - Sport and Spine Rehab, McLean, Virginia
  - Sport and Spine Rehab, Sterling, Virginia